CLINICAL TRIAL: NCT04139031
Title: Corrected Flow Time in the Carotid Artery as a Predictor of Fluid Responsiveness in Mechanically Ventilated Patients With Low Tidal Volume in the Intensive Care Unit
Status: Completed | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2019-0848
Record Dates: First submitted 2019-10-23; First posted 2019-10-25 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Hypovolemic
MeSH Terms: conditions — Hypovolemia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Fluid loading group: Mechanically ventilated patients with low tidal volume in the intensive care unit whom clinician decided to provide fluid for correction of hypovolemia
  Interventions: Device: Ultrasonographic measurement of corrected flow time in carotid artery

INTERVENTIONS:
Device: Ultrasonographic measurement of corrected flow time in carotid artery — Corrected carotid artery flow time is measured using 6-13 MHz linear probe on a portable ultrasound machine. On the two-dimensional image, the optimal image of the long-axis view is obtained at the left common carotid artery. The sample volume is placed on the center of the lumen, 2 cm proximal to the bulb, and a pulsed wave Doppler examination was performed while the Doppler beams were adjusted to ensure < 60° of angle for the best signal. Then, cardiac cycle time and carotid flow time is measured. Carotid flow time is measured between the upstroke of the flow tracing and the dicrotic notch, and it is corrected for pulse rate by dividing flow time by the square root of the cardiac cycle time to calculate corrected carotid artery flow time (flow time/√cycle time).

SUMMARY:
The purpose of this study is to evaluate predictability of carotid corrected flow time for fluid responsiveness in mechanically ventilated patients with low tidal volume in the intensive care unit.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients with age more than 19
2. Undergoing postoperative mechanical ventilation with low tidal volume
3. Clinically diagnosed with hypovolemic status
4. If one of follow criteria is satisfied 1) Systolic blood pressure <90mmHg 2) Mean arterial pressure(MBP)<70mmHg or fall more than 20% from baseline 3) Heart rate >100bpm 4) Urine output <0.5mg/kg/hr more than 1 hour 5) Arterial lactate >2mmol/L 6) Capillary refilling time >3secs

Exclusion Criteria:

1. Body mass index <40 or >15 kg/m2
2. Medical history of carotid artery stenosis >50% or diagnosed while examination
3. Cardiac arrhythmia other than normal sinus rhythm
4. Moderate or severe valvular heart disease, intracardiac shunt, heart failure, pulmonary hypertension
5. Moderate or severe chronic obstructive pulmonary disease
6. Increased intracranial pressure
7. Using vasopressor
8. Pregnancy

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing postoperative mechanical ventilation with low tidal volume
Sampling Method: Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2019-11-05 (Actual); Primary Completion 2020-09-25 (Actual); Study Completion 2020-09-25 (Actual)

PRIMARY OUTCOMES:
Corrected carotid artery flow time during low tidal volume ventilation | Procedure (During low tidal volume ventilation before fluid resuscitation)
  Area under the receiver operating curve of Corrected carotid artery flow time for fluid responsiveness in low tidal volume ventilator setting before fluid resuscitation

SECONDARY OUTCOMES:
Pulse pressure variation during low tidal volume ventilation | Procedure (During low tidal volume ventilation before fluid resuscitation)
  Area under the receiver operating curve of pulse pressure variation for fluid responsiveness in low tidal volume ventilator setting before fluid resuscitation

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Anesthesia and Pain Research Institute, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No